CLINICAL TRIAL: NCT02004821
Title: Génomique de la résistance à la Prise de Poids Dans la Maigreur Constitutionnelle
Brief Title: Clinical Trial in Constitutional Thinness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12.17.NIHS
Record Dates: First submitted 2013-11-15; First posted 2013-12-09 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Individuals With Constitutional Thinness
MeSH Terms: interventions — Proteins; Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renutryl® Booster (Experimental): Renutryl® Booster, an oral nutritional supplement in a 300 ml bottle (600 kcal, 30 g protein, 72 g carbohydrate, 21 g fat).
  Interventions: Dietary Supplement: Renutryl® Booster, an oral nutritional supplement in a 300 ml bottle (600 kcal, 30 g protein, 72 g carbohydrate, 21 g fat). One bottle per day during 14 days.

INTERVENTIONS:
Dietary Supplement: Renutryl® Booster, an oral nutritional supplement in a 300 ml bottle (600 kcal, 30 g protein, 72 g carbohydrate, 21 g fat). One bottle per day during 14 days.

SUMMARY:
The purpose of this study is to evaluate the molecular differences between a group of Constitutionally Thin (CT) subjects and a group of controls.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria specific to subjects with constitutional thinness
* Women: BMI less or equal to 17.5
* Men: BMI less or equal to 18.5
* Stable weight for at least 3 months

Inclusion criteria specific to subjects with normal weight

* Men and women: BMI above or equal to 20 but not more than 25
* Stable weight for at least 3 months
* No previous family history of first or second-degree obesity

Inclusion criteria common to both groups

* Age: between 18 and 35 at the inclusion visit
* Normal blood sugar, liver function, lipid and coagulation profiles
* Signed consent form to participate in the study
* Signed consent form for genetic analysis
* Acceptance of a moderate weight gain of 2 kg (less than 10% of body weight)
* Beneficiary or member of a social security system.

Exclusion Criteria:

* Adults with a legal guardian, or subjects unable to act freely due to a decision by a legal or administrative authority,
* Pregnancy in the case of women
* Women without contraception
* Vegetarian subjects or those with lactose intolerance
* Subjects with an eating disorder (DSM IV)
* Significant alcohol consumption equivalent to more than 10 glasses of wine per week
* Severe progressive disorder (diabetes, for example)
* Subjects who undertake intensive physical activity (more than 3 sessions of physical activity per week)
* Significant tobacco consumption equivalent to more than 10 cigarettes per day
* Depression or psychiatric condition (treated with antidepressant or psychotropic medication), depression questionnaire/score
* Medical or surgical history considered by the investigator to be incompatible with this study (stomach or intestinal surgery, for example)
* Subjects receiving treatment that may interfere with the parameters measured: antihypertensives (blockers, centrally acting antihypertensives), anti-hyperlipidemic agents or corticosteroids for more than 8 days
* Inclusion in a different clinical study within the previous 12 weeks.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Molecular differences (evaluated in plasma, fat and muscle biopsies, urines) between a group of CT subjects and a control group before, during and after 14 days of overnutrition | 6 weeks
  Molecular analyses of plasma, fat and muscle biopsies and urine

SECONDARY OUTCOMES:
Metabolic, anthropometric, histological, and microbiome differences between a group of CT subjects and a control group before, during, and after 14 days of overnutrition | 6 weeks
  * Metabolic differences (eg: lipids, amino-acids… in plasma and urine)
  * Anthropometric differences (eg: weight, BMI, waist/ hip ratio)
  * Histological (eg: muscle and fat tissue biopsies)
  * Inflammation and metabolism specific marker differences
  * Energy metabolism differences (eg: RER, RQ, Cox, Lox…)
  * Bone quality differences (eg: bone mineral density)
  * Microbiome differences

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Estour, Prof., Principal Investigator — CHU de Saint-Étienne
Locations (1):
- CHU de Saint-Étienne, Saint-Etienne, France

REFERENCES:
- [Derived] Cominetti O, Nunez Galindo A, Corthesy J, Carayol J, Germain N, Galusca B, Estour B, Hager J, Gheldof N, Dayon L. Proteomics reveals unique plasma signatures in constitutional thinness. Proteomics Clin Appl. 2022 Sep;16(5):e2100114. doi: 10.1002/prca.202100114. Epub 2022 May 26. PMID 35579096
- [Derived] Bailly M, Germain N, Feasson L, Costes F, Estour B, Hourde C, N Merlet A, Thomas T, Hager J, Pereira B, Thivel D, Courteix D, Galusca B, Verney J. Skeletal muscle of females and males with constitutional thinness: a low intramuscular lipid content and oxidative profile. Appl Physiol Nutr Metab. 2020 Nov;45(11):1287-1298. doi: 10.1139/apnm-2020-0068. Epub 2020 Jun 1. PMID 32479741
- [Derived] Ling Y, Galusca B, Martin FP, Bartova S, Carayol J, Moco S, Epelbaum J, Grouselle D, Boirie Y, Montaurier C, Cuenco J, Minnion JS, Thomas T, Mure S, Hager J, Estour B, Gheldof N, Germain N. Resistance to lean mass gain in constitutional thinness in free-living conditions is not overpassed by overfeeding. J Cachexia Sarcopenia Muscle. 2020 Oct;11(5):1187-1199. doi: 10.1002/jcsm.12572. Epub 2020 Apr 10. PMID 32274897
- [Derived] Ling Y, Carayol J, Galusca B, Canto C, Montaurier C, Matone A, Vassallo I, Minehira K, Alexandre V, Cominetti O, Nunez Galindo A, Corthesy J, Dayon L, Charpagne A, Metairon S, Raymond F, Descombes P, Casteillo F, Peoc'h M, Palaghiu R, Feasson L, Boirie Y, Estour B, Hager J, Germain N, Gheldof N. Persistent low body weight in humans is associated with higher mitochondrial activity in white adipose tissue. Am J Clin Nutr. 2019 Sep 1;110(3):605-616. doi: 10.1093/ajcn/nqz144. PMID 31374571